CLINICAL TRIAL: NCT02010073
Title: A Multicentre, Prospective, Observational, 4-week Inception Cohort Study Being Carried Out by the Acute Respiratory Failure Section of ESICM
Brief Title: Large Observational Study to UNderstand the Global Impact of Severe Acute Respiratory FailurE
Acronym: LUNG-SAFE
Status: Completed | Type: Observational
Sponsor: European Society of Intensive Care Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: LUNG-SAFE
Record Dates: First submitted 2013-11-28; First posted 2013-12-12 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-12

CONDITIONS: Acute Severe Respiratory Failure; Acute Respiratory Distress Syndrome
Keywords: Lung; ARDS; acute; respiratory; syndrome; prognosis; outcome research; respiratory infection; sepsis; organ failure; hypoxaemia
MeSH Terms: conditions — Respiratory Distress Syndrome; Syndrome; Respiratory Tract Infections; Sepsis; Hypoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- One Group: This is a prospective observational study, aimed at collecting an adequate dataset on a large cohort of patients admitted to a large number of ICUs.

SUMMARY:
We wish to prospectively assess the burden of, management and therapeutic approaches to, and outcomes from acute hypoxaemic respiratory failure requiring ventilatory support, during the winter months in both the northern and southern hemispheres. We wish to specifically examine the contribution of ARDS as defined by the Berlin Definition to the burden of hypoxaemic respiratory failure.

Why?

The purpose of this study is to provide new and current data on the disease burden of acute hypoxemic respiratory failure and ARDS. It will answer the following questions:

* What is the frequency and disease burden of acute hypoxaemic respiratory failure in winter?
* What are the aetiologies of acute hypoxaemic respiratory failure requiring ventilatory support?
* What is the incidence of ARDS based on the Berlin definition within this patient cohort?
* What is the mortality from ARDS within this cohort, and how does this vary based on ARDS severity?
* What is the natural history of ARDS?
* What are the key patterns of therapeutic resource utilization, particularly approaches to sustain gas exchange, in these patients?

When?

The study is performed over a 4 week period between February 1st and March 31st 2014 in the Northern Hemisphere and June 1st to August 31st in the Southern Hemisphere.

What data is required?

A basic dataset is collected on all patients admitted with acute acute hypoxaemic respiratory failure requiring ventilatory support, with a more detailed dataset collected on patients diagnosed with ARDS.

DETAILED DESCRIPTION:
In summary, the study will focus on the following items:

* The frequency and disease burden of acute hypoxaemic respiratory failure in winter
* The aetiologies of acute hypoxaemic respiratory failure requiring ventilatory support.
* The incidence of ARDS based on the Berlin definition within this patient cohort
* The mortality from ARDS within this cohort, and how does this vary based on ARDS severity
* Natural history of ARDS (duration and evolution by severity)
* Therapeutic resource utilization

  * Use of treatments, such as recruitment maneuvers, prone positioning, nitric oxide, high frequency oscillation, ECMO, transfer to tertiary hospital from smaller regional ones) according to the severity of the disease
  * Use of non-invasive ventilation in management of ARDS patients (use in different stages: early ARDS versus immediately after extubation).

This is a prospective observational study, aimed at collecting an adequate dataset on a large cohort of patients admitted to a large number of ICUs.

ICUs will be invited to participate on a voluntary basis. ICUs enrolling into existing databases (e.g., ERIC study, ICON audit) will be invited to participate. It is important that participating ICUs commit (by written agreement) to fully comply with the study protocol. ICU recruitment in each country will be spearheaded by a national coordinator Each ICU will be requested to recruit for 4 consecutive 'winter' weeks

1. Northern Hemisphere - 4 week period between February 1st and March 31st 2014.
2. Southern Hemisphere: 4 week period between June 1st - August 31st 2014 There will be 2 data collectors per participating ICU's. Each data collector will undergo an online training program designed to standardize data interpretation [esp. CXR's] and will receive a login authorization following completion of this training.

INCLUSION CRITERIA: All patients admitted to the participating ICUs receiving invasive or noninvasive ventilation will be screened and included in the database.

EXCLUSION CRITERIA: Age < 16.

DATA COLLECTION: Data collection will web based, permitting conditional Data Collection screens, i.e. data collectors will be automatically guided as to which sections to complete based on data entered indicating whether Inclusion Criteria are met. Data collection will be done at 10am each morning. Our aim is to obtain a sample of at least 1000 ARDS patients within the cohort of patients receiving assisted ventilation. The reported incidence of ARDS in ICU patients varies, from 2.2% of ICU admissions develop ARDS in ALIEN, 7.1% in ALIVE Study, to 17.5% of Ventilated patients in KCLIP . A reasonable projection of the incidence of ARDS among patients admitted in ICUs can be estimated to approximate 5% of ICU admission. As a conservative estimate, if a medium-sized ICU admits 50 patients/month and collects data for four, 500 ICUs will be necessary to achieve this number.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the participating ICUs receiving invasive or non-invasive ventilation will be screened and included in the database.

Exclusion Criteria:

* Age < 16

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Our aim is to obtain a sample of at least 1000 ARDS patients within the cohort of patients receiving assisted ventilation.
Sampling Method: Probability Sample
Enrollment: 14000 (Actual)
Dates: Start 2014-02; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Development of ARDS | 28 days

SECONDARY OUTCOMES:
ICU mortality | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: John LAFFEY, MD, Principal Investigator — National University of Galway, Ireland and St Michael's Hospital-University of Toronto, Canada; Antonio PESENTI, MD, Principal Investigator — S Gerardo Hospital, University of Milan-Bicocca, Monza, Italy
Locations (1):
- All Centres Willing to Contribute Are Welcome, Brussels, Belgium

REFERENCES:
- [Derived] Serafini SC, van Meenen DMP, Pisani L, Neto AS, Ball L, de Abreu MG, Algera AG, Azevedo L, Bellani G, Dondorp AM, Fan E, Laffey JG, Pham T, Tschernko EM, Schultz MJ, van der Woude MCE; ERICC; LUNG SAFE; PRoVENT; PRoVENT-iMiC-investigators. Different ventilation intensities among various categories of patients ventilated for reasons other than ARDS--A pooled analysis of 4 observational studies. J Crit Care. 2024 Jun;81:154531. doi: 10.1016/j.jcrc.2024.154531. Epub 2024 Feb 10. PMID 38341938
- [Derived] Amado-Rodriguez L, Rodriguez-Garcia R, Bellani G, Pham T, Fan E, Madotto F, Laffey JG, Albaiceta GM; LUNG SAFE investigators. Mechanical ventilation in patients with cardiogenic pulmonary edema: a sub-analysis of the LUNG SAFE study. J Intensive Care. 2022 Dec 25;10(1):55. doi: 10.1186/s40560-022-00648-x. PMID 36567347
- [Derived] Rezoagli E, McNicholas BA, Madotto F, Pham T, Bellani G, Laffey JG; LUNG SAFE Investigators, the ESICM Trials Group. Presence of comorbidities alters management and worsens outcome of patients with acute respiratory distress syndrome: insights from the LUNG SAFE study. Ann Intensive Care. 2022 May 21;12(1):42. doi: 10.1186/s13613-022-01015-7. PMID 35596885
- [Derived] Madotto F, McNicholas B, Rezoagli E, Pham T, Laffey JG, Bellani G; LUNG SAFE Investigators; ESICM Trials Group. Death in hospital following ICU discharge: insights from the LUNG SAFE study. Crit Care. 2021 Apr 13;25(1):144. doi: 10.1186/s13054-021-03465-0. PMID 33849625
- [Derived] Pham T, Pesenti A, Bellani G, Rubenfeld G, Fan E, Bugedo G, Lorente JA, Fernandes ADV, Van Haren F, Bruhn A, Rios F, Esteban A, Gattinoni L, Larsson A, McAuley DF, Ranieri M, Thompson BT, Wrigge H, Brochard LJ, Laffey JG; LUNG SAFE Investigators and the European Society of Intensive Care Medicine Trials Group. Outcome of acute hypoxaemic respiratory failure: insights from the LUNG SAFE Study. Eur Respir J. 2021 Jun 10;57(6):2003317. doi: 10.1183/13993003.03317-2020. Print 2021 Jun. PMID 33334944
- [Derived] Madotto F, Rezoagli E, Pham T, Schmidt M, McNicholas B, Protti A, Panwar R, Bellani G, Fan E, van Haren F, Brochard L, Laffey JG; LUNG SAFE Investigators and the ESICM Trials Group. Hyperoxemia and excess oxygen use in early acute respiratory distress syndrome: insights from the LUNG SAFE study. Crit Care. 2020 Mar 31;24(1):125. doi: 10.1186/s13054-020-2826-6. PMID 32234077
- [Derived] Duggal A, Rezoagli E, Pham T, McNicholas BA, Fan E, Bellani G, Rubenfeld G, Pesenti AM, Laffey JG; LUNG SAFE Investigators and the ESICM Trials Group. Patterns of Use of Adjunctive Therapies in Patients With Early Moderate to Severe ARDS: Insights From the LUNG SAFE Study. Chest. 2020 Jun;157(6):1497-1505. doi: 10.1016/j.chest.2020.01.041. Epub 2020 Feb 20. PMID 32088180
- [Derived] Boyle AJ, Madotto F, Laffey JG, Bellani G, Pham T, Pesenti A, Thompson BT, O'Kane CM, Deane AM, McAuley DF; LUNG SAFE Investigators; ESICM Trials Group. Identifying associations between diabetes and acute respiratory distress syndrome in patients with acute hypoxemic respiratory failure: an analysis of the LUNG SAFE database. Crit Care. 2018 Oct 27;22(1):268. doi: 10.1186/s13054-018-2158-y. PMID 30367670
- [Derived] Abe T, Madotto F, Pham T, Nagata I, Uchida M, Tamiya N, Kurahashi K, Bellani G, Laffey JG; LUNG-SAFE Investigators and the ESICM Trials Group. Epidemiology and patterns of tracheostomy practice in patients with acute respiratory distress syndrome in ICUs across 50 countries. Crit Care. 2018 Aug 17;22(1):195. doi: 10.1186/s13054-018-2126-6. PMID 30115127
- [Derived] Cortegiani A, Madotto F, Gregoretti C, Bellani G, Laffey JG, Pham T, Van Haren F, Giarratano A, Antonelli M, Pesenti A, Grasselli G; LUNG SAFE Investigators and the ESICM Trials Group. Immunocompromised patients with acute respiratory distress syndrome: secondary analysis of the LUNG SAFE database. Crit Care. 2018 Jun 12;22(1):157. doi: 10.1186/s13054-018-2079-9. PMID 29895331
- [Derived] Madotto F, Pham T, Bellani G, Bos LD, Simonis FD, Fan E, Artigas A, Brochard L, Schultz MJ, Laffey JG; LUNG SAFE Investigators and the ESICM Trials Group. Resolved versus confirmed ARDS after 24 h: insights from the LUNG SAFE study. Intensive Care Med. 2018 May;44(5):564-577. doi: 10.1007/s00134-018-5152-6. Epub 2018 Apr 9. PMID 29632996
- [Derived] de Prost N, Pham T, Carteaux G, Mekontso Dessap A, Brun-Buisson C, Fan E, Bellani G, Laffey J, Mercat A, Brochard L, Maitre B; LUNG SAFE investigators; ESICM trials group; REVA network. Etiologies, diagnostic work-up and outcomes of acute respiratory distress syndrome with no common risk factor: a prospective multicenter study. Ann Intensive Care. 2017 Dec;7(1):69. doi: 10.1186/s13613-017-0281-6. Epub 2017 Jun 19. PMID 28631088
- [Derived] Laffey JG, Madotto F, Bellani G, Pham T, Fan E, Brochard L, Amin P, Arabi Y, Bajwa EK, Bruhn A, Cerny V, Clarkson K, Heunks L, Kurahashi K, Laake JH, Lorente JA, McNamee L, Nin N, Palo JE, Piquilloud L, Qiu H, Jimenez JIS, Esteban A, McAuley DF, van Haren F, Ranieri M, Rubenfeld G, Wrigge H, Slutsky AS, Pesenti A; LUNG SAFE Investigators; ESICM Trials Group. Geo-economic variations in epidemiology, patterns of care, and outcomes in patients with acute respiratory distress syndrome: insights from the LUNG SAFE prospective cohort study. Lancet Respir Med. 2017 Aug;5(8):627-638. doi: 10.1016/S2213-2600(17)30213-8. Epub 2017 Jun 15. PMID 28624388
- [Derived] Laffey JG, Bellani G, Pham T, Fan E, Madotto F, Bajwa EK, Brochard L, Clarkson K, Esteban A, Gattinoni L, van Haren F, Heunks LM, Kurahashi K, Laake JH, Larsson A, McAuley DF, McNamee L, Nin N, Qiu H, Ranieri M, Rubenfeld GD, Thompson BT, Wrigge H, Slutsky AS, Pesenti A; LUNG SAFE Investigators and the ESICM Trials Group. Potentially modifiable factors contributing to outcome from acute respiratory distress syndrome: the LUNG SAFE study. Intensive Care Med. 2016 Dec;42(12):1865-1876. doi: 10.1007/s00134-016-4571-5. Epub 2016 Oct 18. PMID 27757516
- [Derived] Bellani G, Laffey JG, Pham T, Fan E, Brochard L, Esteban A, Gattinoni L, van Haren F, Larsson A, McAuley DF, Ranieri M, Rubenfeld G, Thompson BT, Wrigge H, Slutsky AS, Pesenti A; LUNG SAFE Investigators; ESICM Trials Group. Epidemiology, Patterns of Care, and Mortality for Patients With Acute Respiratory Distress Syndrome in Intensive Care Units in 50 Countries. JAMA. 2016 Feb 23;315(8):788-800. doi: 10.1001/jama.2016.0291. PMID 26903337
- See also: Related Info — http://www.esicm.org/research/LUNG-SAFE